CLINICAL TRIAL: NCT04194905
Title: Bioavailability of a Formulation of Levonorgestrel and Ethinyl Estradiol 0.1 mg/0.02 mg Coated Tablets With Regards to the Marketed Reference Product
Brief Title: Bioavailability of Levonorgestrel/Ethinyl Estradiol Tablets 0.1 mg/0.02 mg With Regards to Reference Product
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Andromaco S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP8814-02; 013-19-V1-080519 (Other: Innolab)
Record Dates: First submitted 2019-11-12; First posted 2019-12-11 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2020-11

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Levonorgestrel; Ethinyl Estradiol; Floors and Floorcoverings; Patents as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levonorgestrel Ethinyl estradiol Test Product (Experimental): Participants will receive two tablets of the test formulation containing Levonorgestrel 0.1 mg and Ethinyl estradiol 0.02 mg. The tablets will be taken with water and in a fasting condition.
  Interventions: Drug: Levonorgestrel 0.1 mg and Ethinyl estradiol 0.02 mg Test Product
- Levonorgestrel Ethinyl estradiol Reference Product (Active Comparator): Participants will receive two tablets of the marketed reference formulation containing Levonorgestrel 0.1 mg and Ethinyl estradiol 0.02 mg. The tablets will be taken with water and in a fasting condition.
  Interventions: Drug: Levonorgestrel 0.1 mg and Ethinyl estradiol 0.02 mg Reference Product

INTERVENTIONS:
Drug: Levonorgestrel 0.1 mg and Ethinyl estradiol 0.02 mg Test Product — Coated Tablets
  Other Names: Investigational Medicinal Product
  Arms: Levonorgestrel Ethinyl estradiol Test Product
Drug: Levonorgestrel 0.1 mg and Ethinyl estradiol 0.02 mg Reference Product — Coated Tablets
  Other Names: Level (Trademark)
  Arms: Levonorgestrel Ethinyl estradiol Reference Product

SUMMARY:
This Pilot study will investigate the bioavailability in fasting women of 2 tablet formulations containing Levonorgestrel 0.1 mg and Ethinyl estradiol 0.02 mg.

The Pilot study will be performed at a single site with 30 subjects. Participants will take 2 tablets of the test product and reference product in 2 periods and 2 sequences (either test after reference or reference after test). There will be a washout of at least 14 days between each study period.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the relative bioavailability of Levonorgestrel and Ethinyl estradiol of 2 tablet formulations with Levonorgestrel 0.1 mg and Ethinyl estradiol 0.02 mg and to demonstrate bioequivalence of both formulations in terms of rate and extent of absorption:

* Test Product: Product manufactured by Laboratorios Andrómaco S.A.
* Reference Product: Level [Trademark], product of Biolab Sanus Farmaceutica Ltda.

The 90% confidence intervals for the intra-subject coefficient of variation (Test versus Reference Product) for the main pharmacokinetic parameters area under the plasma concentration-time curve from time zero to time t (AUC0-t) and from time zero to 72 hours (AUC0-72), and maximum plasma concentration (Cmax) for total Levonorgestrel and Ethinyl estradiol will be determined.

Participants will be confined in the study site for approximately 36 hours during each study period (for 12 hours pre-dosing and for 24 hours post dosing) during which pharmacokinetic (PK) blood samples will be obtained. 16 blood samples will be taken up to 24 hours after the administration in each period. Participants will return to the site to provide additional blood samples at 48 h, and 72 h postdose.

The washout period between the two study periods will be at least 14 days. The samples from each participant will be analyzed with 2 methods of high performance liquid chromatography-tandem mass spectrometry bioanalytical assays to quantify total Levonorgestrel and Ethinyl estradiol in plasma.

The safety objective is to evaluate the tolerability of both formulations in women by collecting adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant and non-breastfeeding women
* Women of childbearing age with an acceptable form of contraception during the study
* 18 to 55 years old inclusive; BMI greater than or equal to 18.51 and less than or equal to 29.99
* Non-smoking or smoke only 3 cigarettes every 7 days
* With results of laboratory tests, electrocardiogram and chest radiography in normal and / or negative or abnormal ranges but without clinical relevance and declared suitable for study by the doctor after the physical examination
* Capable to understand the Informed Consent Form

Exclusion Criteria:

* Study Site staff or family members
* With history of drug and/or alcohol abuse
* Smokers more tan 3 cigarettes every 7 days
* Vitamin supplements intake 7 days prior to the administration of the medications under study
* Any recent change in eating habits or physical exercise
* Using of pharmacological therapy (except over the counter medication use 7 days prior the study)
* Hypersensitivity to the study drug or other related compounds, history of serious adverse reactions or hypersensitivity to any medication
* Use, during 28 days prior to the start of the study, of medications known to alter liver enzyme activity
* Consumption of beverages or food containing grapefruit or pink grapefruit, within 7 days prior to each administration of the study medication and consumption of alcohol, caffeine or beverages or food containing xanthine 24 hours prior each administration of study medication until the last sample of each period
* History of any significant cardiovascular disease
* Acute disease that generates significant physiological changes from the start of the selection until the end of the study
* HIV, Hepatitis B and/or C positive
* Presence or history of thrombophlebitis, thrombosis or thromboembolic disorder, deep vein thrombosis, pulmonary embolism or known coagulopathy.
* Donation or loss of a significant volume (more tan 100 mL) of blood or plasma or platelets during the 3 months prior to the start of the study
* Subjects who have participated in any type of clinical study during the 3 months prior to the start of the study
* History of any gastrointestinal surgery that could affect drug absorption
* Presence of fainting history or fear to blood collection

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-21 (Actual); Primary Completion 2020-11-21 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Total Ethinyl estradiol: area under the plasma concentration-time curve from 0 to 72 hours (AUC0-72) ] | From tablet intake and up to 72 hours after tablet intake
  19 samples up to 72 hours will be taken after the administration in each period.
Total Levonorgestrel: area under the plasma concentration-time curve from 0 to 72 hours (AUC0-72) | From tablet intake and up to 72 hours after tablet intake
  19 samples up to 72 hours will be taken after the administration in each period.
Total Ethinyl estradiol: area under the plasma concentration-time curve from 0 to time t (AUC0-t) | From tablet intake and up to 72 hours after tablet intake
  19 samples up to 72 hours will be taken after the administration in each period.
Total Levonorgestrel: area under the plasma concentration-time curve from 0 to time t (AUC0-t) | From tablet intake and up to 72 hours after tablet intake
  19 samples up to 72 hours will be taken after the administration in each period.
Total Ethinyl estradiol: Maximum plasma concentration (Cmax) | From tablet intake and up to 72 hours after tablet intake
  19 samples up to 72 hours will be taken after the administration in each period. The Cmax will be calculated.
Total Levonorgestrel: Maximum plasma concentration (Cmax) | From tablet intake and up to 72 hours after tablet intake
  19 samples up to 72 hours will be taken after the administration in each period. The Cmax will be calculated.

SECONDARY OUTCOMES:
Total Levonorgestrel: Time to achieve maximum plasma concentration (tmax) | From tablet intake and up to 72 hours after tablet intake
  19 samples up to 72 hours will be taken after the administration in each period. The tmax will be calculated.
Total Ethinyl estradiol: Time to achieve maximum plasma concentration (tmax) | From tablet intake and up to 72 hours after tablet intake
  19 samples up to 72 hours will be taken after the administration in each period. The tmax will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Laboratorios Andromaco, Study Director — Grünenthal Group
Locations (1):
- Innolab, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No